CLINICAL TRIAL: NCT00003194
Title: A Phase I Study of Thiotepa in Combination With Carboplatin and Topotecan With Peripheral Blood Progenitor Cell Support for the Treatment of Children With Recurrent or Refractory Solid Tumors.
Brief Title: Combination Chemotherapy and Peripheral Stem Cell Transplantation in Treating Patients With Recurrent or Refractory Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study enrollment did not meet expected goals
Sponsor: Seattle Children's Hospital (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Doug Hawkins, Investigator, Seattle Children's Hospital
Purpose: Treatment
Other Study IDs: CHMC-6006; CDR0000066029 (Registry Identifier: PDQ (Physician Data Query)); FHCRC-1244.00; NCI-G98-1373
Record Dates: First submitted 2000-04-06; First posted 2003-01-27 (Estimated); Last update posted 2019-04-05 (Actual); Status verified 2019-04

CONDITIONS: Unspecified Childhood Solid Tumor, Protocol Specific
Keywords: unspecified childhood solid tumor, protocol specific
MeSH Terms: interventions — Filgrastim; Carboplatin; Cyclophosphamide; Etoposide; Thiotepa; Topotecan; Peripheral Blood Stem Cell Transplantation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Biological: filgrastim
Drug: carboplatin
Drug: cyclophosphamide
Drug: etoposide
Drug: thiotepa
Drug: topotecan hydrochloride
Procedure: peripheral blood stem cell transplantation

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining chemotherapy with peripheral stem cell transplantation may allow the doctor to give higher doses of chemotherapy drugs and kill more tumor cells.

PURPOSE: Phase I trial to study the effectiveness of combination chemotherapy and peripheral stem cell transplantation in treating patients who have recurrent or refractory solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose of thiotepa in combination with carboplatin and topotecan with peripheral blood stem cell transplantation in patients with recurrent or refractory pediatric solid tumors.
* Determine the toxicity of this regimen in these patients.

OUTLINE: This is a dose escalation study of thiotepa.

Patients may receive 2 courses of mobilization comprising cyclophosphamide and etoposide with filgrastim (G-CSF) support and peripheral blood stem cell (PBSC) collection.

Patients receive thiotepa IV over 2 hours on days 0 and 1; topotecan IV over 30 minutes on days 0-4; and carboplatin IV over 2 hours on days 2 and 3. Patients also receive G-CSF beginning on day 5, 24-36 hours following the last dose of topotecan. PBSC are reinfused on day 6 (36-48 hours following the last dose of topotecan) of each course of therapy. Patients receive 3 courses of therapy.

Cohorts of 3-6 patients receive escalating doses of thiotepa until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose-limiting toxicity.

Patients are followed at 1 and 2 years.

PROJECTED ACCRUAL: A maximum of 24 patients will be accrued into this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven recurrent or refractory pediatric solid tumor
* Bone marrow metastases allowed

PATIENT CHARACTERISTICS:

Age:

* 1 to 30

Performance status:

* 0-2

Life expectancy:

* At least 2 months

Hematopoietic:

* Absolute neutrophil count at least 1,000/mm3
* Platelet count at least 100,000/mm3 (transfusion independent)
* Hemoglobin at least 10 g/dL (RBC transfusion allowed)

Hepatic:

* Bilirubin no greater than 1.5 times normal
* SGOT no greater than 2.5 times normal

Renal:

* Adequate renal function as defined by one of the following:

  * GFR by creatinine clearance
  * Radioisotope GFR
  * Iothalamate at least 70 mL/min

Cardiovascular:

* Adequate cardiac function as defined by one of the following:

  * Ejection fraction at least 55% by MUGA
  * Fractional shortening at least 28% by echocardiogram

Neurologic:

* Adequate CNS function as defined by:

  * Seizure disorder, if present, controlled by anticonvulsants
  * CNS toxicity no greater than grade 2

Other:

* No uncontrolled infections
* Not pregnant or nursing
* No allergy to platinum compounds
* No history of allergy to etoposide (unless mobilization phase not required)

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Recovered from prior immunotherapy
* At least 1 week since prior cytokines
* At least 3 months since prior bone marrow or peripheral blood stem cell transplantation
* No concurrent immunomodulator
* No concurrent cytokines

Chemotherapy:

* At least 3 weeks (6 for nitrosourea) since prior chemotherapy and recovered
* No prior thiotepa
* No other concurrent chemotherapy

Endocrine therapy:

* Not specified

Radiotherapy:

* Recovered from prior radiotherapy
* At least 6 months since prior total body irradiation conditioning
* No concurrent radiotherapy to greater than 10% of total liver, lung, or bone marrow

Surgery:

* Not specified

Ages: 1 Year to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 24 (Estimated)
Dates: Start 1997-07; Primary Completion 2002-12-19 (Actual); Study Completion 2002-12-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Douglas Hawkins, MD, Study Chair — Seattle Children's Hospital
Locations (2):
- United States (2):
  - Children's Hospital and Regional Medical Center - Seattle, Seattle, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington